CLINICAL TRIAL: NCT00626847
Title: Nuclear Genetic and Mitochondrial Influences in Glaucoma
Brief Title: How Does Your Genetic Make-up (Profile) Influence Your Glaucoma?
Status: Completed | Type: Observational
Sponsor: Wills Eye (Other)
Collaborators: Jefferson Medical College of Thomas Jefferson University (Other); Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, George L. Spaeth MD, Director Glaucoma Research Center Wills Eye; Director Medical Research and Education Glaucoma Service Foundation Wills Eye; Esposito Research Professor, Thomas Jefferson University, Wills Eye
Other Study IDs: IRB#07-826
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Primary Open Angle Glaucoma
Keywords: primary open angle glaucoma; Nuclear Genetics; Mitochondrial DNA; POAG
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Primary Open Angle Glaucoma (POAG)
- 2: Controls (Normals, patients without glaucoma)

SUMMARY:
Glaucoma is a group of diseases in which visual loss occurs because of damage to the optic nerve. Research has shown that certain genes may cause glaucoma in some cases. So far, research has only been able to find the genes responsible for glaucoma in a small percentage of people who have glaucoma. The purpose of this project is to study the genes in patients with and without glaucoma to find additional genes that may be responsible for causing glaucoma.

DETAILED DESCRIPTION:
Four tubes of blood will be taken from 100 people. Of those, half will have primary open angle glaucoma (POAG) and the other half will be controls (normals), half will be caucasians and the other half will be african americans, half male and half female. All groups will have a routine ophthalmic eye exam, color vision, snellen vision, and visual field done.

ELIGIBILITY:
Inclusion Criteria:

* 40 yrs
* Caucasian or African American
* Male or female with POAG, PACG, PXFG,
* Normal

Exclusion Criteria:

* Other ophthamic co-morbidities
* Other ethnic groups
* Unable to understand and give informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: glaucoma clinic
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The investigators will quantify the spectrum of changes in mitochondrial respiration, relative mitochondrial DNA content, and oxidative stress associated with different types of glaucoma. | one blood draw

CONTACTS AND LOCATIONS:
Overall Officials: George L Spaeth, MD, Principal Investigator — Wills Eye Institute
Locations (1):
- Wills Eye Glaucoma Service, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Two manuscripts have been written and published.

REFERENCES:
- [Result] Abu-Amero KK, Azad TA, Spaeth GL, Myers J, Katz LJ, Moster M, Bosley TM. Unaltered myocilin expression in the blood of primary open angle glaucoma patients. Mol Vis. 2012;18:1004-9. Epub 2012 Apr 21. PMID 22550394
- [Result] Abu-Amero KK, Azad TA, Spaeth GL, Myers J, Katz LJ, Moster M, Bosley TM. Absence of altered expression of optineurin in primary open angle glaucoma patients. Mol Vis. 2012;18:1421-7. Epub 2012 Jun 1. PMID 22690120